CLINICAL TRIAL: NCT00688142
Title: Magnetoencephalographic Imaging of Sleepiness: The Effect of Armodafinil in Shift Work Sleep Disorder
Brief Title: Sleepiness and Brain Function: The Effect of Armodafinil in Shift Work Sleep Disorder
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Christopher Drake, Ph.D., Henry Ford Health System
Other Study IDs: C10953/6079/ES/US
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Shift Work Sleep Disorder
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Individuals with shift work sleep disorder
- 2: Healthy night shift workers without shift work sleep disorder

SUMMARY:
The investigators hypothesize that in patients with shift work sleep disorder, armodafinil will specifically increase brain activity in the frontal cortex parallel with improvements in deficits of fundamental mechanisms of attention.

DETAILED DESCRIPTION:
The current protocol will utilize a paradigm which is well suited to examine frontal attentional neuronal mechanisms by eliciting event related potential components known to reflect automatic stimulus detection as well as involuntary and voluntary attentional processes. The that end the proposed research has two specific aims. 1) Identify what areas of the frontal lobe and corresponding cognitive functions are impacted by excessive sleepiness in shift work sleep disorder and 2) identify specific brain areas affected by armodafinil and their role in improvement of fundamental attentional processes using a complex cognitive task targeting attentional control.

ELIGIBILITY:
Inclusion Criteria:

* Night shift workers with and without shift work sleep disorder.

Exclusion Criteria:

* Secondary condition to shift work sleep disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population must be healthy night shift workers with a diagnosis of shift work sleep disorder.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Drake, Ph.D., Principal Investigator — Henry Ford Hospital Sleep Disorders & Research Center
Locations (1):
- Henry Ford Hospital Sleep Disorders & Research Center, Detroit, Michigan, United States